CLINICAL TRIAL: NCT00694343
Title: Evaluation of the Efficacy of 6% Hydroxyethyl Starch (HES, 130/0.4) in Normal Saline Compared to Ringer's Lactate Solution for the Prevention of Hypotension During Spinal Anesthesia for Cesarean Section
Brief Title: Efficacy of Voluven® for the Prevention of Hypotension During Spinal Anesthesia for Cesarean Section
Acronym: CAESAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-HE06-03; EudraCT no.:2007-006065-32
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Hypotension
Keywords: Cesarean section; spinal anesthesia; hypotension
MeSH Terms: conditions — Hypotension | interventions — Hydroxyethyl Starch Derivatives; Sodium Chloride; Solutions; HES 130-0.4; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): 500 mL of HES 130/0.4 (6%) and 500 mL Ringer's Lactate Solution
  Interventions: Drug: HES 130/0.4 (6%) in sodium chloride (solution for infusion)
- Group B (Active Comparator): 1000 mL Ringer's Lactate solution
  Interventions: Drug: Ringer's Lactate solution

INTERVENTIONS:
Drug: HES 130/0.4 (6%) in sodium chloride (solution for infusion) — 500 mL of HES 130/0.4 (6%) and 500 mL Ringer's Lactate Solution
  Other Names: Voluven®
  Arms: Group A
Drug: Ringer's Lactate solution — 1000 mL Ringer's Lactate solution
  Other Names: Ringer's Lactate
  Arms: Group B

SUMMARY:
The aim of the study is to evaluate the efficacy of Voluven® in the prevention of maternal hypotension in women undergoing spinal anesthesia for cesarean section

DETAILED DESCRIPTION:
Intravenous fluid administration prior to spinal anesthesia for cesarean section is an established part of anesthetic practice for the prevention of maternal hypotension. Systematic reviews of clinical data suggest the usefulness of administering colloids to decrease the incidence of hypotension This study will compare the clinical efficacy and safety of HES 130/0.4 (6%) in normal saline vs. Ringer's lactate solution in prevention of hypotension during spinal anesthesia for elective cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean section applying spinal anesthesia
* ≥ week 37 of gestation
* Singleton pregnancy

Exclusion Criteria:

* Suspicion of any hypertensive disease
* Parturient in labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | Time between induction of spinal anesthesia until delivery

SECONDARY OUTCOMES:
Minimum of systolic blood pressure until delivery | between induction of anesthesia and delivery
Maternal heart rate between induction of anesthesia and delivery | between induction of anesthesia and delivery
Onset and duration of hypotension between induction of anesthesia and delivery | between induction of anesthesia and delivery
Phenylephrine requirements to keep systolic blood pressure equal or higher than 95% of baseline value | between induction of anesthesia and delivery

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Mercier, Professor, Principal Investigator — Hôpital Béclère, Service Anesthésie-Réanimation, 157 Rue de la Porte de Trivaux, 92140 Clamart, France
Locations (14):
- France (14):
  - CHU Clermont Ferrand - Hotel Dieu, Service Anesthesie-Reanimation, Clermont-Ferrand
  - Höpital Louis-Mourier - Service d'Anesthesie, Colombes
  - Département d'Anesthésie-Réanimation - Centre Hospitalo-Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Hopital Jeanne de Flandre, CHU, Lille
  - CHU Hotel Dieu, Service Anesthesie, Lyon
  - Hopital Arnaud de Villeneuve - Service Anesthésie-Réanimation, Montpellier
  - Hopital de l'Archet, Service Anesthesie-Reanimation, Nice
  - Hopital Caremeau, CHU, Service Anesthesie, Nîmes
  - Hopital Cochin, Service Anesthesie-Reanimation Chirurgicale, Paris
  - Hôpital Armand-Trousseau, Service d'anesthésie-réanimation, Paris
  - Hopital Robert Debre, CHU, Service Anesthesie, Reims
  - Hopital Hautepierre, CHU, Service Reanimation Chirurgicale, Strasbourg
  - Hopital Foch,Service Anesthesie, Suresnes
  - Unité d'anesthésie - Maternité Paule de Viguier, Toulouse

REFERENCES:
- [Derived] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD002251. doi: 10.1002/14651858.CD002251.pub4. PMID 32619039
- [Derived] Mercier FJ, Diemunsch P, Ducloy-Bouthors AS, Mignon A, Fischler M, Malinovsky JM, Bolandard F, Aya AG, Raucoules-Aime M, Chassard D, Keita H, Rigouzzo A, Le Gouez A; CAESAR Working Group. 6% Hydroxyethyl starch (130/0.4) vs Ringer's lactate preloading before spinal anaesthesia for Caesarean delivery: the randomized, double-blind, multicentre CAESAR trial. Br J Anaesth. 2014 Sep;113(3):459-67. doi: 10.1093/bja/aeu103. Epub 2014 Jun 26. PMID 24970272